CLINICAL TRIAL: NCT01935869
Title: Combined Cumulative Irritation Potential and Repeat Insult Patch Test of LEO 90100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: LP0053-66
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-07

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LEO 90100 (Experimental)
  Interventions: Drug: LEO 90100
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle
- Petrolatum ointment (Other)
  Interventions: Drug: Petrolatum ointment

INTERVENTIONS:
Drug: LEO 90100
  Arms: LEO 90100
Drug: Vehicle
  Arms: Vehicle
Drug: Petrolatum ointment
  Arms: Petrolatum ointment

SUMMARY:
The purpose of this study is to determine the skin irritation potential and sensitisation potential of LEO 90100 and the vehicle after repeated applications on the skin of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Following verbal and written information about the trial, subject must provide signed and dated informed consent before any study related activities are carried out.
* 2. Healthy male or female subjects, 18 to 65 years of age inclusive at screening.

Exclusion Criteria:

* 1. Female subjects who are pregnant, of childbearing potential and who wish to become pregnant during the study, or who are breast feeding
* 2. Subjects with any systemic or cutaneous disorder that might interfere with the evaluation of the test site reactions (e.g. atopic dermatitis, contact eczema, psoriasis) 3. Subjects with scars, moles or other abnormal pigmentation of the skin or skin type that could, in any way, confound interpretation of the study results (skin type V and VI on the Fitzpatrick scale)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mean Cumulative Irritation index and maximal dermal response during induction phase | 3 weeks
Number of subjects with positive sensitisation reaction at each test site in the challenge phase | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- CPCAD, Centre de Pharmacologie Clinique Appliquée à la Dermatologie, Hôpital de l'Archet 2, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Queille-Roussel C, Liljedahl M, Clonier F, Lacour JP. Phase I evaluation of the dermal safety of the fixed combination calcipotriene plus betamethasone dipropionate aerosol foam and foam vehicle. J Am Acad Dermatol. 2015:72 Suppl 1;AB211 (P844).
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en